CLINICAL TRIAL: NCT03205280
Title: Assessment of a Clinical Decision Support System (CADIMS) for Improving Multiple Sclerosis Diagnostic Accuracy
Brief Title: Clinical Decision Support System (CADIMS) for MS Diagnostic
Acronym: POCADIMS
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Collaborators: Association Neuro-Bretagne (Unknown); Institut National de Recherche en Informatique et en Automatique (Other); Groupement de Coopération Sanitaire e-Santé Bretagne (Unknown); Institut de Recherche Technologique b<>com (Unknown)
Responsible Party: Sponsor
Other Study IDs: 35RC16_8968 POCADIMS
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2018-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis, Relapsing-Remitting, Computer-Assisted Diagnosis, MRI, Diagnosis, Treatment Efficacy
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Background The results obtained in clinical research led to a new paradigm for the treatment of patients affected with multiple sclerosis (MS): "no evidence of disease activity". This means having each patient monitored with high quality imaging. To this purpose, researchers have developed segmentation algorithms for automated reading of MRIs, facilitating longitudinal comparisons, and allowing an accurate assessment of the number and the volume of focal lesions. We have thus a powerful strategic biomarker for the treatment of MS.

   Due to the relevance of comparing over time the evolution of lesions (lesion load) and brain atrophy, the French Society of Neuroradiology edited standardized national recommendations. The MS French Observatory (OFSEP) has adopted these recommendations, in order to harmonize exams for all patients all over the country. At an international level as well, MRI have been put at the heart of the therapeutic strategy.

   Therefore, we need now to create the conditions able to implement, collect and analyze imaging data according to these recommendations.

   This is the meaning of the MUSIC project, which aims to develop and assess a standardized monitoring MRI control tool for therapeutic decision.

   CADIMS is this tool. It is based on an integration of several segmentation algorithms developed by INRIA and an image viewer developed by b<>com and included in a regional images-sharing server ETIAM Nexus. This tool is a help showing segmented brain T2 lesions, gadolinium-enhanced T1 lesions and news T2 lesions appeared from the previous MRI exam, in a multicenter clinical context.
2. Objective To evaluate the accuracy of MS lesions detection on cerebral MRI by comparing the CADIMS tool to the expert consensus.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years-old
* Patient with relapsing-remitting multiple sclerosis, according to the 2010 Mc Donald's criteria
* EDSS<4
* Disease duration < 10 years
* To insure a clinical demand of 2 brain MRIs within 12 months of the installation of an immunomodulatory therapy
* MRI brain scanner acquired according to the OFSEP recommendations installation of an immunomodulatory therapy

Exclusion Criteria:

* Progressive MS
* no consent of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Relapsing-remitting multiple sclerosis patients
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Concordance among the number of new T2 lesions, the total number of T2 lesions and the number of gadolinium enhanced lesions on brain MRIs identified by the CADIMS tool and by the expert consensus | At the end of the enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe FERRE, PhD, Principal Investigator — Rennes University Hospital
Locations (5):
- France (5):
  - Centre Hospitalier Bretagne Sud, Lorient
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Centre Hospitalier, Rennes
  - Centre d'imagerie médicale de la découverte, St-Malo
  - Centre Hospitalier Bretagne Atlantique, Vannes